CLINICAL TRIAL: NCT06247475
Title: Generating Fast and Slow for Entree Level Medical Knowledge
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taiwan Emergency Medical Technician Association (Unknown)
Responsible Party: Sponsor
Other Study IDs: 202308059RINB
Record Dates: First submitted 2024-01-29; First posted 2024-02-08 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-01

CONDITIONS: Patient Satisfaction
Keywords: Artificial Intelligence; Decision Making, Shared
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Medical professionals: Attending physicians of National Taiwan University Hospital
  Interventions: Other: Answers generated by ChatGPT
- Healthcare-related professionals: Medical Radiation Technologist of National Taiwan University Hospital
  Interventions: Other: Answers generated by ChatGPT
- Medical students: Medical students of National Taiwan University College of Medicine who have passed the first stage of Taiwan Medical Licencing Exam.
  Interventions: Other: Answers generated by ChatGPT
- General public: Volunteers from Taiwan Emergency Medical Technician Association
  Interventions: Other: Answers generated by ChatGPT

INTERVENTIONS:
Other: Answers generated by ChatGPT — Participants will assign a satisfaction score based on the appropriateness of each answer.

SUMMARY:
The generative artificial intelligence tool, ChatGPT, has garnered widespread interest since its launch. This innovative multimedia platform has the potential to enhance medical communication and health education, thereby improving medical accessibility and reducing the burden on healthcare professionals. Some studies have indicated that ChatGPT achieves higher levels of satisfaction in counseling compared to human healthcare professionals. Additionally, research has shown that ChatGPT's performance in answering objective structured clinical examination questions is comparable to that of typical medical students. However, in both scenarios, it still requires editing by professionals before being used. Moreover, a recent meta-analysis evaluating ChatGPT's ability in various types of medical exams revealed inconsistent results. Before its application and actual integration into clinical practice, the investigators need to comprehend the advantages, disadvantages, and relevant limitations of ChatGPT in the field of medical communication. This study aims to simulate virtual consultations between ChatGPT, acting as a health professional, and study participants, serving as patients. It will evaluate the participants' satisfaction with the virtual consultation questions, categorized by different levels of cognition through Bloom's Taxonomy. This study plans to recruit medical professionals, healthcare-related professionals, medical students from National Taiwan University Hospital, and the general public. Two researchers will select 20 questions from the USMLE step 3 practice tests and the second stage of the Taiwan Medical Licensing Examination. These questions will be categorized into different levels of cognition based on knowledge, comprehension, application, analysis, synthesis, or evaluation. ChatGPT 3.5 and 4.0 will answer these 20 questions without specifying the question's level of cognition. Each participant will review the answers to these 20 questions and assign a satisfaction score based on the appropriateness of each answer.

ELIGIBILITY:
Inclusion Criteria:

1. National Taiwan University Hospital

   * Medical professionals
   * Healthcare-related professionals
   * Medical students
2. Taiwan Emergency Medical Technician Association.

   * Volunteers

Exclusion Criteria:

* N/A.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The medical professionals, healthcare-related professionals, and medical students refer to attending physician, medical radiation technologist from National Taiwan University Hospital, and medical students from National Taiwan University College of Medicine, respectively. The general public refer to volunteers from Taiwan Emergency Medical Technician Association.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between satisfaction and Bloom's taxonomy | baseline (at completion of study questionnaire)
  Divided by the four participant groups

SECONDARY OUTCOMES:
Correctness of answers | baseline (at completion of study questionnaire)
  Answers from ChatGPT 3.5/4.0 and the answers provided by Medical Licencing Exam institutions

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Data would be shared by request.